CLINICAL TRIAL: NCT00651183
Title: Non-motor Symptoms (Depressive Symptoms) of Parkinson's Disease and Their Course Under Pramipexole Treatment
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.649
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Pramipexole immediate release

SUMMARY:
The objective of this PMS study is the evaluation of depressive symptoms measured with Unified Parkinson's Disease Rating Scale (UPDRS) Part I (mentation, behavior and mood) and with Hospital Anxiety and Depression Scale Depression Subscore (HADS-D) under pramipexole treatment in early and advanced PD patients. In addition it will be investigated whether improvement of depressive symptoms is linked to improvement in motor function (UPDRS Part III). 250 patients diagnosed with Parkinson's disease (PD) will be investigated by 80 specialists (neurologists or neurologists/psychiatrists) across Austria. Pramipexole will be taken orally at an initial dosage of 0.375 mg/day (using a three times daily schedule independently of food intake) and can be titrated upwards, as required, at weekly intervals to a maximum total daily dose of 4,5 mg (TID) as per Summary of Product Characteristics (SPC).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD with or without fluctuations
* Indication for treatment with Pramipexole
* Presence of at least mild depressive symptoms (as judged by the treating physician)
* Ability to reliably complete a self-rating scale (Hospital Anxiety and Depression Scale (HADS))

Exclusion Criteria:

* Any contraindications according to the Summary of Product Characteristics (SPC), hypersensitivity to pramipexole or to any of the excipients
* Ongoing treatment with pramipexole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (57):
- Austria (57):
  - Boehringer Ingelheim Investigational Site, Amstetten
  - Boehringer Ingelheim Investigational Site, Bad Hall
  - Boehringer Ingelheim Investigational Site, Bad Ischl
  - Boehringer Ingelheim Investigational Site, Bad Radkersburg
  - Boehringer Ingelheim Investigational Site, Baden
  - Boehringer Ingelheim Investigational Site, Bregenz
  - Boehringer Ingelheim Investigational Site, Bruck an der Mur
  - Boehringer Ingelheim Investigational Site, Deutschlandsberg
  - Boehringer Ingelheim Investigational Site, Dornbirn
  - Boehringer Ingelheim Investigational Site, Eisenstadt
  - Boehringer Ingelheim Investigational Site, Feldkirch
  - Boehringer Ingelheim Investigational Site, Feldkirchen in Kärnten
  - Boehringer Ingelheim Investigational Site, Gänserndorf
  - Boehringer Ingelheim Investigational Site, Gmunden
  - Boehringer Ingelheim Investigational Site, Graz
  - Boehringer Ingelheim Investigational Site, Grieskirchen
  - Boehringer Ingelheim Investigational Site, Hall in Tirol
  - Boehringer Ingelheim Investigational Site, Hallein
  - Boehringer Ingelheim Investigational Site, Hermagor
  - Boehringer Ingelheim Investigational Site, Hohenems
  - Boehringer Ingelheim Investigational Site, Hollabrunn
  - Boehringer Ingelheim Investigational Site, Horn
  - Boehringer Ingelheim Investigational Site, Imst
  - Boehringer Ingelheim Investigational Site, Innsbruck
  - Boehringer Ingelheim Investigational Site, Judenburg
  - Boehringer Ingelheim Investigational Site, Kapfenberg
  - Boehringer Ingelheim Investigational Site, Klagenfurt
  - Boehringer Ingelheim Investigational Site, Klosterneuburg
  - Boehringer Ingelheim Investigational Site, Knittelfeld
  - Boehringer Ingelheim Investigational Site, Krems
  - Boehringer Ingelheim Investigational Site, Kufstein
  - Boehringer Ingelheim Investigational Site, Leoben
  - Boehringer Ingelheim Investigational Site, Lienz
  - Boehringer Ingelheim Investigational Site, Lilienfeld
  - Boehringer Ingelheim Investigational Site, Linz
  - Boehringer Ingelheim Investigational Site, Melk
  - Boehringer Ingelheim Investigational Site, Neunkirchen
  - Boehringer Ingelheim Investigational Site, Oberwart
  - Boehringer Ingelheim Investigational Site, Ried im Innkreis
  - Boehringer Ingelheim Investigational Site, Salzburg
  - Boehringer Ingelheim Investigational Site, Sankt Pölten
  - Boehringer Ingelheim Investigational Site, Sankt Veit an der Glan
  - Boehringer Ingelheim Investigational Site, Scheibbs
  - Boehringer Ingelheim Investigational Site, Schwechat
  - Boehringer Ingelheim Investigational Site, Spital An Der Drau
  - Boehringer Ingelheim Investigational Site, St Johann im Pongau
  - Boehringer Ingelheim Investigational Site, Stegersbach
  - Boehringer Ingelheim Investigational Site, Stockerau
  - Boehringer Ingelheim Investigational Site, Telfs
  - Boehringer Ingelheim Investigational Site, Traun
  - Boehringer Ingelheim Investigational Site, Vienna
  - Boehringer Ingelheim Investigational Site, Villach
  - Boehringer Ingelheim Investigational Site, Vöcklabruck
  - Boehringer Ingelheim Investigational Site, W. Neustadt
  - Boehringer Ingelheim Investigational Site, Wels
  - Boehringer Ingelheim Investigational Site, Wolfsberg
  - Boehringer Ingelheim Investigational Site, Wörgl

RESULTS

PARTICIPANT FLOW:
Groups:
- Early (PD): Early Parkinson's Disease (PD) patients
- Advanced PD: Advanced Parkinson's Disease (PD) patients
Period: Overall Study
Arm/Group | Early (PD) | Advanced PD
Started | 189 (For one patient the information was not given, therefore, the patient was listed "missing") | 97
Completed | 169 (Case Report Form (CRF) listed reasons for early termination, of which one was) | 87 ("other reasons". No explanation was required to be given by the physicians)
Not Completed | 20 | 10
Not completed — Lack of Efficacy | 1 | 0
Not completed — Efficacy insufficient + patients wish | 0 | 1
Not completed — Tolerability insufficient | 5 | 2
Not completed — Tolerability insufficient +Patients wish | 0 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Other reasons | 4 | 2
Not completed — missing | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety set (SAF)
Groups:
- Early PD: Early Parkinson's Disease (PD) patients
- Total: Total of all reporting groups
Arm/Group | Early PD | Advanced PD | Total
Number analyzed (Participants) | 189 | 97 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline data are presented for the safety analysis set (including data of all 286 patients - 189 early PD patients / 97 advanced PD patients - reported to have received at least one dose of study drug, i.e. pramipexole). For Age, Continuous the number of patients with age information collected was 187 for Early PD and 94 for Advanced PD.
  years | 69.1 (9.44) | 73.8 (6.97) | 70.6 (8.96)
Sex/Gender, Customized [Number; unit: participants] — Baseline data are presented for the safety analysis set (including data of all 286 patients - 189 early PD patients / 97 advanced PD patients - reported to have received at least one dose of study drug, i.e. pramipexole).
  For two patients the participating physicians did not enter the gender in the CRF, therefore, they were listed as "missing"
  participants
    Female | 80 | 35 | 115
    Male | 108 | 61 | 169
    missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part I (Mentation, Behaviour and Mood)
Description: Rating scale scored from 0 (none) - 4 (severe). The UPDRS Part I (Mentation, Behaviour and Mood during the Past Week) consist of 4 items, each of them is scored from 0 (normal) to 4 (severe). Reduction in this score over time is interpreted as improvement.
  Total UPDRS part I score ranges from 0 = best score to 16 = worst score
Time Frame: Baseline and Final (visit 3) - Change from baseline (i.e. decrease of score)
Population: Only those patients of the full analysis set (FAS) with an evaluation of UPDRS Part I at visit 3 were included in this analysis
Measure: Median (Inter-Quartile Range); unit: Points on a scale
Arm/Group | Early PD | Advanced PD
Number analyzed (Participants) | 165 | 85
Points on a scale | 2 [1.00 to 3.00] | 2 [1.00 to 3.00]

2. Primary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale - HADS-D Depression Subscore
Description: Depression Scale - 7 items scored for each individual question from 0 = best and 3 = worst.
  HADS is a self-assessment scale for the symptom severity of anxiety disorders and depression.
  It comprises of 14 items, thereof seven statements describe anxiety and seven statements depression. Each answer is rated on a four-point scale (0-3). All seven answers are summarized and calculated to a total score to the anxiety scale and to the depression scale with a maximum score of 21 points for each scale.
Time Frame: Baseline and Final (visit 3) - Change from baseline (i.e. decrease of score)
Population: Only those patients of the full analysis set (FAS) with an evaluation of HADS-D at visit 3 were included in this analysis
Measure: Median (Inter-Quartile Range); unit: Points on a scale
Arm/Group | Early PD | Advanced PD
Number analyzed (Participants) | 161 | 79
Points on a scale | 3 [1.00 to 6.00] | 4 [2.00 to 7.00]

3. Primary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale - HADS-A Anxiety Subscore
Description: Anxiety Scale - 7 items scored for each individual question from 0 = best and 3 = worst.
  HADS is a self-assessment scale for the symptom severity of anxiety disorders and depression.
  It comprises of 14 items, thereof seven statements describe anxiety and seven statements depression. Each answer is rated on a four-point scale (0-3). All seven answers are summarized and calculated to a total score to the anxiety scale and to the depression scale with a maximum score of 21 points for each scale.
Time Frame: Baseline and Final (visit 3) - Change from baseline (i.e. decrease of score)
Population: Only those patients of the full analysis set (FAS) with an evaluation of HADS-A at visit 3 were included in this analysis
Measure: Median (Inter-Quartile Range); unit: Points on a scale
Arm/Group | Early PD | Advanced PD
Number analyzed (Participants) | 161 | 79
Points on a scale | 2 [1.00 to 4.00] | 4 [1.00 to 6.00]

4. Primary Outcome: Change From Baseline in UPDRS Part III (Motor Examination)
Description: 14 components rating scale with 27 items scored by 0 (none) - 4 (severe)
Time Frame: Baseline and Final (visit 3) - Change from baseline (i.e. decrease of score)
Population: Only those patients of the full analysis set (FAS) with an evaluation of UPDRS Part III at visit 3 were included in this analysis
Measure: Median (Inter-Quartile Range); unit: Points on a scale
Arm/Group | Early PD | Advanced PD
Number analyzed (Participants) | 172 | 87
Points on a scale | 9 [4.00 to 14.00] | 10 [6.00 to 17.00]

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: The safety analysis set (SAF) includes the data of all 286 patients (189 early PD patients/ 97 advanced PD patients - reported to have received at least one dose of study drug, i.e. pramipexole
Arm/Group | Early PD | Advanced PD
Serious Adverse Events (participants affected / at risk) | 0/189 | 1/97
Other Adverse Events (participants affected / at risk) | 0/189 | 0/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early PD (N=189) | Advanced PD (N=97)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.